CLINICAL TRIAL: NCT01979601
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenously Administered LGT209 in Healthy Volunteers and Patients With Hypercholesterolemia on Stable Doses of Statin Medications
Brief Title: Safety, Tolerability, PK and PD of LGT209 in Healthy Volunteers and Patients With Hypercholesterolemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLGT209X2101
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia,; LGT209,; PCSK9,; LDL-C
MeSH Terms: conditions — Hypercholesterolemia; Hypercholesterolemia, Autosomal Dominant, 3

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (12):
- Patient: LGT209 0.3 mg/kg (Experimental): 0.3 mg/kg LGT209 intravenous administration in patients on stable doses of statins
  Interventions: Drug: LGT209
- Patient: LGT209 1 mg/kg (Experimental): 1 mg/kg LGT209 intravenous administration in patients on stable doses of statins
  Interventions: Drug: LGT209
- Patient: LGT209 3 mg/kg (Experimental): 3 mg/kg LGT209 intravenous administration in patients on stable doses of statins
  Interventions: Drug: LGT209
- Patient: LGT209 10 mg/kg (Experimental): 10 mg/kg LGT209 intravenous administration in patients on stable doses of statins
  Interventions: Drug: LGT209
- Patient: LGT209 20 mg/kg (Experimental): 20 mg/kg LGT209 intravenous administration in patients on stable doses of statins
  Interventions: Drug: LGT209
- Healthy Volunteers: LGT209 0.3 mg/kg (Experimental): 0.3 mg/kg LGT209 intravenous administration in healthy volunteers
  Interventions: Drug: LGT209
- Healthy Volunteers: LGT209 1 mg/kg (Experimental): 1 mg/kg LGT209 intravenous administration in healthy volunteers
  Interventions: Drug: LGT209
- Healthy Volunteers: LGT209 3 mg/kg (Experimental): 3 mg/kg LGT209 intravenous administration in healthy volunteers
  Interventions: Drug: LGT209
- Healthy Volunteers: LGT209 10 mg/kg (Experimental): 10 mg/kg LGT209 intravenous administration in healthy volunteers
  Interventions: Drug: LGT209
- Healthy Volunteers: 20 mg/kg (Experimental): 20 mg/kg LGT209 intravenous administration in healthy volunteers
  Interventions: Drug: LGT209
- Patient: Placebo (Placebo Comparator): Matching intravenous placebo in patients on stable doses of statins
  Interventions: Drug: Placebo
- Healthy Volunteers: Placebo (Placebo Comparator): Matching intravenous placebo in healthy volunteers
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LGT209 — 150 mg lyophilized powder in glass vial
  Arms: Healthy Volunteers: 20 mg/kg; Healthy Volunteers: LGT209 0.3 mg/kg; Healthy Volunteers: LGT209 1 mg/kg; Healthy Volunteers: LGT209 10 mg/kg; Healthy Volunteers: LGT209 3 mg/kg; Patient: LGT209 0.3 mg/kg; Patient: LGT209 1 mg/kg; Patient: LGT209 10 mg/kg; Patient: LGT209 20 mg/kg; Patient: LGT209 3 mg/kg
Drug: Placebo — Placebo comparator
  Arms: Healthy Volunteers: Placebo; Patient: Placebo

SUMMARY:
This study is designed to measure the effects of LGT209 when given intravenously to patients with high cholesterol who are on stable doses of statin medications, and to healthy subjects with elevated cholesterol

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers: Male and female subjects 18 to 70 years of age, in general good health but with high cholesterol
* Statin patients: Male and female patients 18 to 70 years of age, with high cholesterol on stable statin therapy for at least 3 months

Exclusion Criteria:

* Healthy volunteers: History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes
* Women of child-bearing potential unless using highly effective methods of contraception
* Statin patients: Use of any prescription drugs for lipid lowering other than HMG CO-A reductase inhibitors (statins); use of two concurrent antihypertensive medications is allowed, provided stable dosing has been achieved for the prior 3 months
* Women of child-bearing potential unless using highly effective methods of contraception

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events, serious adverse events and death | from Screening until Day 141
Change from baseline in low density lipoprotein-cholesterol (LDL-C) concentration in healthy volunteers | Baseline, Day 29
  Baseline was defined as the arithmetic mean of all the pre-treatment values (i.e. Screening, Day -1 and predose on Day 1)
Change from baseline in proprotein convertase subtilisin/kexin type 9 (PCSK9) in healthy volunteers | Baseline, Day 29
  Baseline was defined as the arithmetic mean of all the pre-treatment values (i.e. Screening, Day -1 and predose on Day 1)
Pharmacokinetics of LGT209: : Area under the serum concentration-time curve from time zero to infinity (AUC0-inf) of LGT209 in patients and healthy volunteers following intravenous administration | Day 1 (1, 2, 4, 6, 8, 12 hrs post dose); Post-dose at 24 hr (Day 2); 48 hr (Day 3), 96 hr (Day 5), Days 8, 11, 15, 22, 29, 43, 57, 71, 85, 113, 141
Pharmacokinetics of LGT209: observed maximum serum concentrations (Cmax) of LGT209 in patients and healthy volunteers following intravenous administration | Day 1 (1, 2, 4, 6, 8, 12 hrs post dose); Post-dose at 24 hr (Day 2) 48 hr (Day 3), 96 hr (Day 5), Days 8, 11, 15, 22, 29, 43, 57, 71, 85, 113, 141
Pharmacokinetics of LGT209: Area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration (AUC0-last) of LGT209 in patients and healthy volunteers following intravenous administration | Day 1 (1, 2, 4, 6, 8, 12 hrs post dose); Post-dose at 24 hr (Day 2) 48 hr (Day 3), 96 hr (Day 5), Days 8, 11, 15, 22, 29, 43, 57, 71, 85, 113, 141
Pharmacokinetics of LGT209: Elimination half-life associated with the terminal slope of a semi-logarithmic concentration-time curve (T1/2) of LGT209 in patients and healthy volunteers following intravenous administration | Day 1 (1, 2, 4, 6, 8, 12 hrs post dose); Post-dose at 24 hr (Day 2) 48 hr (Day 3), 96 hr (Day 5), Days 8, 11, 15, 22, 29, 43, 57, 71, 85, 113, 141
Number of healthy volunteers with adverse events, serious adverse events and death | from Screening until Day 141

SECONDARY OUTCOMES:
Pharmacokinetics of intravenous LGT209 in relationship to concentrations of PCSK9 and LDL-C in patients and healthy volunteers | Day 1 (1, 2, 4, 6, 8, 12 hrs post dose); Post-dose at 24 hr (Day 2) 48 hr (Day 3), 96 hr (Day 5), Days 8, 11, 15, 22, 29, 43, 57, 71, 85, 113, 141
Change from baseline in low density lipoprotein-cholesterol (LDL-C) concentration in patients | Baseline, Day 29
  Baseline was defined as the arithmetic mean of all the pre-treatment values (i.e. Screening, Day -1 and predose on Day 1)
Change from baseline in proprotein convertase subtilisin/kexin type 9 (PCSK9) in patients | Baseline, Day 29
  Baseline was defined as the arithmetic mean of all the pre-treatment values (i.e. Screening, Day -1 and predose on Day 1)
Pharmacokinetics of LGT209: Area under the serum concentration-time curve from time zero to time 't' (AUC0-t) | Day 1 (1, 2, 4, 6, 8, 12 hrs post dose); Post-dose at 24 hr (Day 2) 48 hr (Day 3), 96 hr (Day 5), Days 8, 11, 15, 22, 29, 43, 57, 71, 85, 113, 141
  In AUC 0-t, t is a defined as time point after administration of LGT209 in patients and healthy volunteers following intravenous administration
Pharmacokinetics of LGT209: Dose-normalized area under the serum concentration-time curve (AUC/D) of LGT209 in patients and healthy volunteers following intravenous administration | Day 1 (1, 2, 4, 6, 8, 12 hrs post dose); Post-dose at 24 hr (Day 2) 48 hr (Day 3), 96 hr (Day 5), Days 8, 11, 15, 22, 29, 43, 57, 71, 85, 113, 141
Pharmacokinetics of LGT209: Dose-normalized maximum serum concentrations (Cmax/D) of LGT209 in patients and healthy volunteers following intravenous administration | Day 1 ( 1, 2, 4, 6, 8, 12 hrs post dose); Post-dose at 24 hr (Day 2) 48 hr (Day 3), 96 hr (Day 5), Days 8, 11, 15, 22, 29, 43, 57, 71, 85, 113, 141
Pharmacokinetics of LGT209: Volume of distribution during the terminal elimination phase (Vz) of LGT209 in patients and healthy volunteers following intravenous administration | Day 1 (1, 2, 4, 6, 8, 12 hrs post dose); Post-dose at 24 hr (Day 2) 48 hr (Day 3), 96 hr (Day 5), Days 8, 11, 15, 22, 29, 43, 57, 71, 85, 113, 141
Pharmacokinetics of LGT209: Volume of distribution at steady state (Vss) of LGT209 in patients and healthy volunteers following intravenous administration | Day 1 (1, 2, 4, 6, 8, 12 hrs post dose); Post-dose at 24 hr (Day 2) 48 hr (Day 3), 96 hr (Day 5), Days 8, 11, 15, 22, 29, 43, 57, 71, 85, 113, 141
Pharmacokinetics of LGT209: Mean residence time (MRT) of LGT209 in patients and healthy volunteers following intravenous administration | Day 1 (1, 2, 4, 6, 8, 12 hrs post dose); Post-dose at 24 hr (Day 2) 48 hr (Day 3), 96 hr (Day 5), Days 8, 11, 15, 22, 29, 43, 57, 71, 85, 113, 141
Pharmacokinetics of LGT209: the systemic (or total body) clearance from serum following intravenous administration | Day 1 (1, 2, 4, 6, 8, 12 hrs post dose); Post-dose at 24 hr (Day 2) 48 hr (Day 3), 96 hr (Day 5), Days 8, 11, 15, 22, 29, 43, 57, 71, 85, 113, 141

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - Novartis Investigative Site, Miami Gardens, Florida
  - Novartis Investigative Site, Fargo, North Dakota